CLINICAL TRIAL: NCT07133581
Title: Design, Development, and Validation of FEXO: A Playful-Recreational Exercise Intervention for Institutionalized Frail Older Adults to Improve Intrinsic Functional and Cognitive Capacity: A Randomized Controlled Trial
Brief Title: Design and Validation of FEXO: A Playful Exercise Program for Institutionalized Frail Older Adults
Acronym: FEXO-FRAIL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-98
Record Dates: First submitted 2025-07-25; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Frailty Syndrome; Sarcopenia
Keywords: frailty; sarcopenia; intrinsic capacity; Institutionalized older adults; playful exercise; multicomponent exercise
MeSH Terms: conditions — Frailty; Sarcopenia | interventions — Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wait-List Control Group (No Intervention): Participants in this group will continue their usual daily activities for 14 weeks without receiving the FEXO intervention. After this period, they will be offered the same 14-week FEXO program as the experimental group, following the same structure, supervision, and exercise content.
- FEXO Multicomponent Playful Exercise (Experimental): Participants in this group will follow the FEXO program, a 14-week multicomponent playful-recreational exercise intervention. The program includes 3 supervised sessions per week (55-60 minutes each) and incorporates aerobic, resistance, balance, flexibility, and gait exercises delivered in a playful group-based format using motivational materials. The 14-week program is structured into an initial 2-week familiarization phase followed by three progressive 4-week levels. Exercises are adapted and progressively intensified according to individual capacity.
  Interventions: Other: FEXO (Fun Exercise for Older Adults)

INTERVENTIONS:
Other: FEXO (Fun Exercise for Older Adults) — A 14-week supervised multicomponent playful exercise program for institutionalized older adults. It consists of 3 sessions per week (55-60 minutes), including aerobic, strength, balance, flexibility, and gait exercises in a group-based, game-like setting. The structure includes 2 weeks of familiarization followed by 3 progressive 4-week levels. The intervention aims to improve intrinsic capacity, reduce frailty, and enhance physical and cognitive function.
  Arms: FEXO Multicomponent Playful Exercise

SUMMARY:
This multicenter randomized controlled trial aims to evaluate the effectiveness of a playful multicomponent exercise intervention (FEXO - Fun Exercise for Older Adults) on intrinsic capacity, frailty, and functional health in institutionalized older adults aged over 75. The FEXO program combines aerobic, strength, balance, and flexibility training in a recreational format. Participants will be randomized to an experimental group (receiving the 14-week FEXO program) or a wait-list control group (continuing daily routines). After the first intervention phase, the control group will also complete the program. Primary outcomes include improvements in intrinsic capacity domains (cognition, locomotion, vitality, sensory, and psychological), frailty phenotype (Fried criteria), and physical function.

DETAILED DESCRIPTION:
Frailty is a dynamic syndrome marked by diminished physiological reserves and increased vulnerability to stressors. It is prevalent among institutionalized older adults and is associated with higher risks of dependency, hospitalization, and reduced quality of life. Evidence shows that physical inactivity and sedentary behavior significantly contribute to the onset and progression of frailty, especially in long-term care settings.

The World Health Organization (WHO) introduced the concept of Intrinsic Capacity in 2015, emphasizing a multidimensional view of healthy aging that includes cognition, mobility, vitality, sensory function, and psychological well-being. Preserving or enhancing intrinsic capacity is critical to prolonging independence and life quality among older adults.

This trial assesses the effectiveness of the FEXO program, a playful multicomponent exercise intervention designed to enhance intrinsic capacity and reduce frailty in adults over 75 years of age residing in geriatric care centers of the Ballesol Group (Valencia and Alicante). The intervention combines aerobic, strength, balance, gait, and flexibility exercises delivered in a recreational and group-based format using playful tools (e.g., foam balls, scarves, bubbles). Participants will engage in three 55-60 minute sessions per week over 14 weeks.

The study follows a wait-list controlled randomized design. Participants will be randomized to one of two groups: (1) the experimental group, which receives the FEXO intervention immediately, and (2) the control group, which continues routine activities during the first 14 weeks, followed by delayed participation in the program. Outcomes will be measured at baseline (T0), post-intervention (T1, at 14 weeks), and follow-up (T2, 28 weeks post-baseline for the control group).

Primary and secondary outcomes include: Fried's Frailty Phenotype, Short Physical Performance Battery (SPPB), Timed Up and Go Test (TUG), grip strength (JAMAR), walking speed (10-MWT), cognitive status (MMSE), nutritional status (MNA), depressive symptoms (GDS, CSDD), balance (Berg Balance Scale), and quality of life indicators.

This trial responds to the need for evidence-based interventions in institutionalized elderly populations, supporting WHO guidelines for healthy aging and promoting holistic care by integrating physical activity into daily routines through enjoyable, motivating formats.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥75 years.
* Resident in a long-term care facility (residencia geriátrica) affiliated with the Ballesol group (Levante area: Valencia and Alicante).
* Provide informed consent (or consent by legal representative, if appropriate).
* Functional and/or cognitive status that allows them to participate in basic physical activity and understand and follow basic verbal instructions.

Exclusion Criteria:

* Unstable medical condition or uncontrolled chronic disease.
* Severe cognitive impairment or advanced dementia that prevents comprehension or adherence to the intervention, determined by clinical assessment or MMSE <15.
* Severe physical disability.
* Active infectious disease or acute condition requiring isolation or rest.
* Participation in another structured physical activity or rehabilitation program during the study period.
* End-of-life situation or terminal illness.
* Any condition that, in the judgment of the research or clinical team, would interfere with participation or data collection.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2025-09-04 (Estimated); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intrinsic Capacity (IC) | Before and inmediately after the intervention
  This composite outcome evaluates changes in intrinsic capacity, following the five-domain model proposed by the World Health Organization: cognition, vitality, locomotion (function), sensory function, and psychological well-being. Each domain is assessed through one standardized test: the Mini-Mental State Examination (MMSE) for cognition, the Mini Nutritional Assessment (MNA) for vitality, the Short Physical Performance Battery (SPPB) for locomotion, self-reported vision and hearing for sensory function, and the Cornell Scale for Depression in Dementia (CSDD) for psychological well-being. Each test contributes up to a maximum of 2 points, according to predefined cut-off values. For the cognitive domain (MMSE), 2 points are assigned if ≥27, 1 point if 10-26, and 0 points if 0-9. For vitality (MNA), 2 points are assigned if 24-30, 1 point if 17-23, and 0 points if <17. For locomotion (SPPB), 2 points are assigned if ≥10, 1 point if 3-9, and 0 points if 0-2. For sensory function (self-r
Frailty (Fried's Phenotype) | Before and inmediately after the intervention
  Frailty status will be assessed using Fried's phenotype, which classifies participants as robust (0 criteria), pre-frail (1-2 criteria), or frail (3-5 criteria) based on five components: unintentional weight loss, exhaustion, low physical activity, slow gait speed, and weak grip strength. Improvement is defined as transition to a lower frailty category (e.g., from frail to pre-frail).

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Before and inmediately after the intervention
  The SPPB evaluates lower-extremity function through three subtests: standing balance (performed with feet together, semi-tandem, and tandem), gait speed over a 4-meter distance, and a five-times sit-to-stand test. Each subtest is scored from 0 to 4, for a total score ranging from 0 to 12. Higher scores indicate better physical performance. The SPPB is predictive of disability, hospitalization, and mortality in older adults.
Timed Up and Go Test (TUG) | Before and inmediately after the intervention
  This test assesses functional mobility and risk of falling. Participants are instructed to rise from a standard chair, walk 3 meters, turn around, walk back, and sit down. The total time (in seconds) is recorded. Lower times indicate better mobility and balance. The TUG has high predictive value for fall risk in frail older populations.
Grip Strength (JAMAR Dynamometer) | Before and inmediately after the intervention
  Grip strength will be measured using a JAMAR hand dynamometer, with participants seated, the elbow at 90°, forearm in a neutral position, and wrist slightly extended. The best of three trials is recorded in kilograms. Grip strength is a core indicator of sarcopenia and a strong predictor of functional decline, morbidity, and mortality. Higher values reflect better upper-limb muscle strength.
10-Meter Walk Test (10-MWT) | Before and inmediately after the intervention
  Participants will perform two walking trials over 10 meters: one at habitual pace and one at maximum pace. The time to walk the central 6-meter portion is recorded and converted into meters per second (m/s). Gait speed is a validated marker of frailty, physical function, and fall risk. Higher walking speeds reflect better functional status.
Mini-Mental State Examination (MMSE) | Before and inmediately after the intervention
  The MMSE evaluates general cognitive status through domains including orientation, memory, attention, language, and visuospatial skills. It yields a score from 0 to 30, with higher scores indicating better cognitive function. It is widely used for screening and monitoring cognitive impairment in older adults.
Mini Nutritional Assessment (MNA) | Before and inmediately after the intervention
  The MNA is a validated tool for detecting malnutrition or risk of malnutrition in older adults. It includes 18 items covering anthropometry, general health, dietary intake, and subjective assessment. Total scores range from 0 to 30: scores ≥24 indicate normal nutrition, 17-23.5 suggest risk of malnutrition, and <17 indicate malnutrition. Higher scores reflect better nutritional status.
Geriatric Depression Scale (GDS) | Before and inmediately after the intervention
  The GDS short form (15 items) will be used to screen for depressive symptoms in participants. Responses are binary (yes/no), and total scores are calculated. Higher scores indicate more depressive symptoms; scores >5 may indicate clinical depression. Lower scores represent better psychological well-being.
Berg Balance Scale (BBS) | Before and inmediately after the intervention
  This 14-item scale assesses balance and postural control in older adults. Each task (e.g., standing, reaching, turning) is scored from 0 (unable) to 4 (independent), with a total score ranging from 0 to 56. Scores below 45 suggest increased fall risk. Higher scores reflect better balance.
Barthel Index | Before and inmediately after the intervention
  This scale measures independence in 10 basic activities of daily living (ADLs), including feeding, grooming, bathing, dressing, bowel and bladder control, toilet use, transfers, mobility, and stair use. Scores range from 0 to 100, with higher scores indicating greater functional independence. The index is commonly used in geriatric and rehabilitation settings.
Cornell Scale for Depression in Dementia | Before and inmediately after the intervention
  The Cornell Scale for Depression in Dementia (CSDD) will be used to assess depressive symptoms in participants with or without cognitive impairment. The scale consists of 19 items covering mood-related signs, behavioral disturbances, physical signs, cyclic functions, and ideational disturbances. Each item is rated from 0 to 2 (0 = absent, 1 = mild or intermittent, 2 = severe), based on interviews with both the patient and an informant. Total scores range from 0 to 38, with higher scores indicating more severe depressive symptoms. Scores above 10 suggest probable major depression, while scores above 18 are highly indicative of a depressive disorder. Lower scores represent better psychological well-being.
Self-reported Vision | Before and inmediately after the intervention
  Self-reported vision will be assessed through a single-item question asking participants to rate their visual ability. Responses are scored as follows: 0 = severe difficulty or complete blindness, 0.5 = mild to moderate difficulty, and 1 = no difficulty. Higher scores indicate better sensory function.
Self-reported Hearing | Before and inmediately after the intervention
  Self-reported hearing will be assessed through a single-item question asking participants to rate their hearing ability. Responses are scored as follows: 0 = severe difficulty or complete deafness, 0.5 = mild to moderate difficulty, and 1 = no difficulty. Higher scores indicate better sensory function.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Lisón Párraga, Dr, Principal Investigator — Cardenal Herrera University

IPD SHARING:
Plan to Share IPD: Undecided